CLINICAL TRIAL: NCT01468012
Title: Imaging the Neurobiology of Behavioral and Medication Treatment for Cocaine Dependence
Acronym: COST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6022; 6022 (Other: NYSPI IRB)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; levodopa; carbidopa; entacapone
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — carbidopa, levodopa drug combination; entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levodopa carbidopa and entacapone (LCE) (Experimental): 400mg/100mg/200mg, twice daily dosing of levodopa carbidopa and entacapone (LCE)
  Interventions: Drug: levodopa carbidopa and entacapone (LCE)
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levodopa carbidopa and entacapone (LCE) — 400mg/100mg/200mg, twice daily
  Arms: levodopa carbidopa and entacapone (LCE)
Drug: Placebo — matched placebo for LCE condition dosed twice daily
  Arms: Placebo

SUMMARY:
The proposed study will look at cocaine dependent individuals and will consist of three consecutive phases: 1) the 2-week outpatient lead-in phase during which behavioral therapy will be administered; 2) the 15-21 day inpatient phase (during which participants will start study medication of levodopa,carbidopa and entacapone (LCE) and will undergo brain imaging and 3) the 24 weeks outpatient treatment trial. The purpose is to see if treatment with LCE may reverse baseline brain deficits and if this change is associated with clinical improvement. Hypothesis is that treatment with LCE, compared to placebo, increases abstinence from cocaine over a 12-week trial in combination with behavioral treatment with voucher incentives.

DETAILED DESCRIPTION:
Cocaine dependence remains a serious public health problem; however no clearly effective pharmacological treatments have been identified to date. The investigators hypothesize that identification of subgroups of cocaine-dependent patients will help to develop targeted and more effective treatments. The investigators have observed that 30-40% of cocaine-dependent patients who enter our medication trials achieve abstinence during the lead-in period (the two weeks prior to starting medication). Initial abstinence is strongly predictive of abstinence during the subsequent medication trial. The investigators have also observed that a low dopamine release in the striatum is associated with greater choice of cocaine in volunteers and failure of cocaine-dependent patients to respond to behavioral treatment. The investigators hypothesize that individuals who have difficulties in achieving abstinence have a deficit in dopaminergic functioning and correcting this deficit using dopaminergic medication LCE (levodopa in combination with carbidopa and entacapone) will result in clinical improvement.

The proposed study will consist of three consecutive phases: 1) the 2-week outpatient lead-in phase during which behavioral therapy will be administered; 2) the 15-21 day inpatient phase (during which participants will start study medication and will undergo brain imaging; one PET and two fMRI scan sessions); and 3) the 24 weeks outpatient treatment trial.

Study medication (LCE or placebo) will be administered in a double-blind, placebo controlled manner for one week during inpatient phase followed by 12 weeks of the outpatient trial. During the remaining 12 weeks of the outpatient trial participants will receive therapy only.

The purpose of the lead-in phase is to identify patients who do not achieve abstinence in response to behavioral treatment. Subsequently, two matched subgroups of participants (half who achieved abstinence and half who did not achieve abstinence) will undergo the [11C] raclopride displacement PET brain imaging procedure. This procedure allows the measurement of dopamine release in response to a single dose of methylphenidate, and the investigators will determine if failure to achieve abstinence during the lead-in period is associated low dopamine transmission.

All participants in the proposed study will also undergo a functional MRI with the Motivational Incentive Delay task (fMRI/MID). This task is thought to reflect dopaminergic transmission in the brain-reward system but is safer and more feasible than PET. The investigators hypothesize that fMRI/MID will correlate strongly with results from the PET procedure, thereby suggesting that it also reflects the status of striatal dopamine functioning. In addition, a group of healthy controls will undergo one fMRI scan in order to validate the procedure and to assess if a deficit can be detected in cocaine-dependent participants. Cocaine-dependent participants will undergo two fMRI/MID, one at baseline and another after a week of treatment with LCE to assess if treatment with LCE may reverse baseline deficits and if this change is associated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 21-50.
* Meets DSM-IV criteria for current cocaine dependence, supported by a positive urine for cocaine metabolites
* Voluntarily seeking treatment for cocaine dependence
* Absence of other medical or psychiatric disorders that are unstable and would interfere with participation.
* Absence of any suspicious skin changes, suggestive of melanoma, during the full body exam
* Able to give informed consent.

Exclusion Criteria:

* Current DSM-IV criteria of other substance use disorders with the exception of nicotine dependence, and mild to moderate alcohol or cannabis abuse or dependence. Alcohol or cannabis abuse or dependence may be included provided that cocaine is the predominant problem, and medical detoxification is not indicated; alcohol and cannabis use are common among cocaine dependent patients and their categorical exclusion would impede recruitment and result in a sample of limited generalizability; secondary analyses will explore whether they exert any moderating effects on the main findings.
* Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV organic mental disorder, psychotic disorder, bipolar disorder, recurrent severe MDD, OCD, or eating disorder. Participants with depressive disorder (provided that the score on the Hamilton Depression Scale is less than 20) and those with ADHD symptoms may be included, since these are common, often reflect effects of chronic drug use, and may improve with behavioral treatment and cessation or reduction of drug use.
* Unstable medical disorders, or medical disorders that might interfere with study participation, including seizure disorder.
* Significant current suicidal risk or 1 or more suicide attempts within the past year
* Concurrent treatment with psychotropic medications
* Positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control
* Baseline systolic BP of > 140 and < 100, diastolic BP > 90 and < 60 and baseline HR greater than 90.
* Any clinically significant heart abnormality or cardiovascular disease
* History of glaucoma
* History of melanoma or current suspicious undiagnosed skin lesions
* History of allergic reaction or adverse reaction to study medications (levodopa/carbidopa/entacapone; methylphenidate; raclopride).
* Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" by Shellock
* Lifetime exposure to radiation in the workplace, or history of participation in nuclear medicine procedures, including research protocols
* Individuals who are predominantly left handed. Based on a score <50 on the Edinburg Handed Inventory (E.H.I.).

Inclusion Criteria(fMRI study-healthy controls):

* Adult, age 21-50.
* No current DSM-IV psychiatric or substance use disorders
* Absence of other medical disorders that are unstable and would interfere with participation.
* Able to give informed consent.

Exclusion Criteria (fMRI study-healthy controls):

* Current or recent DSM-IV psychiatric or substance use disorders
* Past history of any major Axis I disorder (e.g., psychotic disorders, bipolar disorder, recurrent major depressive disorder, OCD or eating disorders).
* Unstable medical disorders, or medical disorders that might interfere with study participation.
* Concurrent treatment with psychotropic medications
* Positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control *
* Baseline systolic BP of > 140 and < 100, diastolic BP > 90 and < 60 and baseline HR greater than 90.
* Any clinically significant heart abnormality or cardiovascular disease
* History of allergic reaction or adverse reaction to study medications (methylphenidate; raclopride).
* Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" by Shellock
* Individuals who are predominantly left handed. Based on a score <50 on the Edinburg Handed Inventory (E.H.I.).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levodopa Carbidopa and Entacapone (LCE) | Placebo | Non-randomized
Started | 9 | 10 | 4
Completed | 7 | 9 | 0
Not Completed | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levodopa Carbidopa and Entacapone (LCE) | Placebo | Non-randomized | Total
Number analyzed (Participants) | 9 | 10 | 4 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 4 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 7 | 10 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 4 | 20
  White | 0 | 0 | 0 | 0
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Urine Toxicology
Description: Abstinence will be assessed by urine toxicology results collected 3x/week during the 24 week trial or for the length of participation
Time Frame: collected 3x/week for 24 weeks of trial or for the duration of the participants involvement in the study.
Population: Urine toxicology results were not collected
Arm/Group | Levodopa Carbidopa and Entacapone (LCE) | Placebo | Non-randomized
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Retention in Treatment
Description: The number of participants who completed the 12-week medication phase of the study.
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Non-randomized: Participants who dropped from the study prior to randomization
Arm/Group | Levodopa Carbidopa and Entacapone (LCE) | Placebo | Non-randomized
Number analyzed (Participants) | 9 | 10 | 4
participants | 7 | 9 | 0

ADVERSE EVENTS:
Arm/Group | Levodopa Carbidopa and Entacapone (LCE) | Placebo | Non-randomized
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10 | 0/4
Other Adverse Events (participants affected / at risk) | 3/9 | 5/10 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa Carbidopa and Entacapone (LCE) (N=9) | Placebo (N=10) | Non-randomized (N=4)
Hospitalization for leg numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The participant was hospitalized for numbness and pain in the left leg which occurred in the non-medication follow-up phase of the study. The participant was diagnosed with Multiple Sclerosis during the hospitalization
Hospitalization for shortness of breath (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — It was determined that the participant had a presence of Sinus of Valsalva aneurysm on Aortic Valve.
Hospitalization for Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The participant was hospitalized for numbness and pain in the left leg which occurred in the non-medication follow-up phase of the study. The participant was diagnosed with Multiple Sclerosis during the hospitalization
Hospitalization for chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — It was determined that the participant had a presence of Sinus of Valsalva aneurysm on Aortic Valve.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa Carbidopa and Entacapone (LCE) (N=9) | Placebo (N=10) | Non-randomized (N=4)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0)
Orthostatis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
increased libido (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Increased appetite (General disorders) | 1 (1) | 0 (0) | 0 (0)
GI Upset (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prolonged Erection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Irregular Heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No